CLINICAL TRIAL: NCT03575728
Title: Telemetry-Triggered Educational Content Delivery Using MyChart in Mood Disorders
Brief Title: Delivering Telemetry-Triggered Educational Content Using MyChart in Mood Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. David Kreindler, MD, Sunnybrook Health Sciences Centre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0382017
Record Dates: First submitted 2018-06-21; First posted 2018-07-02 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Bipolar Disorder; Mood Disorders
Keywords: Mental Health; Information Technology; Chronic Disease Prevention and Management; Support Patient Self-Care
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Based on self-report answers to screening questions, participants will be divided into two groups: (i) those who screen positive for a history of mood disorders and (ii) all other participants. All outcome measures apply only to the mood disorder group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mood disorder (Other): Participants who screen positive for a history of mood disorders
  Interventions: Other: MyChart-MHT
- Other (Other): Participants who do not screen positive for a history of mood disorders
  Interventions: Other: MyChart-MHT

INTERVENTIONS:
Other: MyChart-MHT — All participants in this study will receive targeted psycho-educational interventions from time to time based on symptom severity reports as determined by the software algorithm

SUMMARY:
Mood disorders - principally major depressive disorder and bipolar disorder - are a significant public health issue affecting one in four people during their lives in total, over 8 million Canadians are affected by mood disorders, costing the economy over $6 billion annually. At Sunnybrook, 75% of inpatient mental health admissions are due to mood disorders. Mood disorders are generally recurrent: approximately half of depression is recurrent; chronic bipolar disorder is typical. Use of ratings scales by patients and clinicians to track symptoms has also been shown to enhance outcomes such as remission, medication adherence, and patient engagement. Education is considered a key component of treating mood disorders. However, which educational information is useful can vary: in depression, changes in illness severity have been shown to affect what information is absorbed, and timing is also important.To address this, this project will deliver, for the first time ever, a system for using data from patients with mood disorders' electronic mood journals, integrated into Sunnybrook's "MyChart" personal health record system, to drive just-in-time delivery of educational interventions, using feedback from users to maximize its usefulness.

DETAILED DESCRIPTION:
This project will integrate mood-journaling software ("MHT") developed here at Sunnybrook (SHSC) into SHSC's "MyChart" patient portal system. Next, using alternating expert input and input from focus groups of patients, we will develop a library of educational content and rules to select and drive delivery of content that will, for the first time, allow patients with mood disorders to receive customized, just-in-time educational content using their own self-report data to drive selection and timing of the delivery of the content. While we expect that this innovation should be beneficial to its users, we cannot assess this without adequate numbers of users. So, in this project, we will make this system available to MyChart users for six months and collect ongoing feedback on user satisfaction, continuously refining the system over the six months with the goal of steadily increasing the number of users frequently using this system.

ELIGIBILITY:
Inclusion Criteria:

i) Registered user of Sunnybrook Health Sciences Centre "MyChart" electronic patient portal

Exclusion Criteria:

-

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Utilization rate | Six month period of study
  Trend in utilization rate over time in users in 'mood disorder' arm

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada